CLINICAL TRIAL: NCT05882773
Title: Asian Myeloproliferative Neoplasm (MPN) Registry - An Asian Myeloid Working Group (AMWG) Project.
Brief Title: Asian Myeloproliferative Neoplasm (MPN) Registry
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: AMWG002
Record Dates: First submitted 2023-05-21; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Myeloproliferative Neoplasm; Polycythemia Vera; Essential Thrombocythemia; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis; Primary Myelofibrosis; Primary Myelofibrosis, Prefibrotic Stage; Primary Myelofibrosis, Fibrotic Stage
Keywords: Myeloproliferative neoplasm; Epidemiology; Outcome; Prognostic factors
MeSH Terms: conditions — Myeloproliferative Disorders; Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Peripheral blood and bone marrow aspirate
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multinational, multicenter, prospective and retrospective, observational, cohort study of patients with myeloproliferative neoplasm.

DETAILED DESCRIPTION:
This is a multinational, multicenter, prospective and retrospective, observational, cohort registry of patients with MPN. The registry mainly involves study centres in Asia including but not limited to Hong Kong, Singapore, Malaysia, Taiwan, Korea and Thailand. Clinicopathologic characteristics, cytogenetic characteristics, mutational characteristics, treatment characteristics, outcomes and survivals of Asian patients MPN diagnosed between 2010-2025 will be collected to establish clinical registry.

Data on the clinicopathologic characteristics, cytogenetics, mutational profile, prognostic scoring treatment characteristics, responses to treatment, outcome and survivals will be collected through routine clinic visits and/or reviewing medical records. Data will be collected at diagnosis, and approximately every 6 months thereafter (for prospective data) and at progression until death/study termination.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old at the time of diagnosis of MPN.
2. Subject was diagnosed with one of the following disorders according to the 2017 WHO classification (for patients diagnosed before 2017, the bone marrow reports will be re-evaluated according to the 2017 WHO classification):

   1. Polycythaemia vera
   2. Essential thrombocythemia
   3. Primary myelofibrosis, pre-fibrotic/early stage
   4. Primary myelofibrosis, overt fibrotic stage
   5. Post-polycythaemia vera myelofibrosis
   6. Post-essential thrombocythaemia myelofibrosis
   7. MPN-unclassifiable
3. All subjects need to provide informed consent.

Exclusion Criteria:

A subject will not be eligible if he/she meets any of the following criteria:

1. Subject was diagnosed with myelodysplastic syndrome, myelodysplastic syndrome/myeloproliferative neoplasm, or chronic myeloid leukaemia BCR-ABL1 positive, under the 2017 WHO classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three study cohorts will be involved in the study. They are:
  Prospective cohort - Subjects will be enrolled in the study at their diagnosis of MPN. All data will be collected on-study prospectively.
  Partial prospective/retrospective cohort (partial-P/R) - Subjects will be enrolled in the study after they have been diagnosed of MPN for a period of time and still being followed up clinically (alive). Data from study enrollment forward will be collected prospectively at around 6-month intervals on-study. Data prior to study enrollment are the events of interest happened and will be collected retrospectively.
  Retrospective cohort - Subjects enrolled in the study after they were diagnosed of MPN and died/lost to follow. All data will be collected retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time to progression to secondary myelofibrosis (for PV and ET) | 10 years
  Measured in months, from date of diagnosis of MPN to date of documentation of secondary myelofibrosis (event), death (event) or latest follow-up (censor). Patient without an event will be censored at date last known to be progression-free
Progression-free survival (PFS) | 10 years
  Measured in months, from date of diagnosis of MPN to the date of the first MDS or AML or death due to any cause. Patient without an event will be censored at date last known to be progression-free and alive.
Overall survival (OS) | 10 years
  Measured in months from the date of diagnosis of MDS until the date of death due to any cause. Patient who is alive will be censored at the date last known alive

CONTACTS AND LOCATIONS:
Overall Officials: Harinder Gill, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Medicine, Queen Mary Hospital, Hong Kong, Hong Kong